CLINICAL TRIAL: NCT01671683
Title: A Phase II Study of Additional Four-week Chemotherapy With Capecitabine During the Resting Periods After Six-week Neoadjuvant Chemoradiotherapy in Patients With Locally Advanced Rectal Cancer
Brief Title: Additional Chemotherapy After Neoadjuvant Chemoradiotherapy in Patients With Locally Advanced Rectal Cancer
Status: Completed | Type: Observational
Sponsor: Chungnam National University (Other)
Responsible Party: Principal Investigator, Ji Yeon Kim, Associate Professor, Chungnam National University
Other Study IDs: CNUH 10
Record Dates: First submitted 2012-08-21; First posted 2012-08-23 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-08

CONDITIONS: Rectal Cancer
Keywords: rectal cancer; neoadjuvant chemoradiotherapy; Capecitabine
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of additional neoadjuvant chemotherapy with capecitabine during the resting periods in patients with locally advanced rectal cancer.

DETAILED DESCRIPTION:
Neoadjuvant chemoradiotherapy (NCRT) has been used as standard treatment modality in patients with locally advanced rectal cancer (LARC) because of increased local control, enhanced sphincter preservation, and less toxicity.NCRT has enhanced down-staging of tumor and reduced local recurrence. However, survival benefit of NCRT has not been demonstrated and the rate of distant metastasis was still reported as high as 30%.

Patients with pathologic complete remission (pCR) after NCRT have shown excellent survival benefit. We inferred that additional chemotherapy during the resting period could enhance the pCR rate. The aim of the present study is to evaluate the safety and efficacy of an additional 4-week chemotherapy with capecitabine after the conventional 6-week NCRT in patients with LARC.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven, locally advanced adenocarcinoma of the rectum
* an Eastern Cooperative Oncology Group (ECOG) score of 0-2
* adequate function of major organs
* a signed informed consent.

Exclusion Criteria:

* other co-existing malignancy or malignancy within the last 5 years prior to enrollment
* severe concurrent medical or psychiatric disorders
* prior RT to pelvis
* pregnant or lactating patients

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients of our hospital
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2010-07; Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ji Yeon Kim, MD., PhD, Principal Investigator — Surgical Oncology Research Lab
Locations (1):
- Chungnam National University Hospital, Daejeon, South Korea